CLINICAL TRIAL: NCT06480617
Title: The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Brief Title: Observational, Bivariate Analysis of Clinical Big Data in Patients With Cervical Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-KY347
Record Dates: First submitted 2024-06-25; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Progression-free Survival Was Defined From Date of Surgery to Disease Progression Post-surgery or Death or Last Follow-up; Overall Survival Was Defined as Time From Surgery to Death From Any Cause or Last Follow-up
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LNM(+): Postoperative pathology suggests lymph node metastasis
- LNM(-): Postoperative pathology did not suggest lymph node metastasis

SUMMARY:
This is a large non-interventional observational bidirectional study planned to collect clinically relevant data and prognostic follow-up information of patients with cervical cancer who were seen at our center from 2010.01.01 to the end of this study.

DETAILED DESCRIPTION:
This study is a large-scale observational, bi-directional analytical study, which collects clinical data from patients with cervical cancer who have received treatment in the Department of Gynecologic Oncology of the First Hospital Affiliated to the University of Science and Technology of China (Anhui Provincial Hospital), including age, weight, BMI, menopausal status, history of the current disease, past history, specialized examinations, results of tests, results of genetic testing, pathology-related data, and information related to surgery, etc. The diagnosis, subsequent treatment, and follow-up of the subjects follow the routine clinical procedures of the clinical center. The diagnosis and subsequent treatment and follow-up of the subjects followed the routine clinical procedures of the clinical center, and the follow-up data of the enrolled patients were collected every six months: imaging, tumor markers, recurrence and treatment. And clinical big data analysis. Therefore, patients who meet the enrollment criteria can be included, and the sample size is based on the actual number of cases included.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. patients with a clear pathological diagnosis of cervical cancer;
3. all patients included in this study were diagnosed after 1 January 2010
4. Diagnosis or treatment of cervical cancer at the centres covered by this study;
5. exemption from informed consent or signing of an informed consent form.

Exclusion Criteria:

1. Loss of contact during the follow-up period for no apparent reason;
2. Discharged from the hospital for follow-up treatment at an outside institution with unknown treatment status;
3. The investigator considers the patient unsuitable for participation in this study;
4. cases where the clinical diagnosis is in doubt or unclear.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cervical cancer patients seen and treated at the Department of Gynaecological Oncology of the First Affiliated Hospital of the University of Science and Technology of China (Anhui Provincial Hospital)
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 5 years

SECONDARY OUTCOMES:
overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yin Zhou, MD, Study Chair — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Locations (1):
- Anhui Provincal Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No